CLINICAL TRIAL: NCT05438875
Title: The Combination of ATRA and Eltrombopag as the Treatment Strategy for Glucocorticoid-Resistant/Relapsed ITP Based on the Stratification of the New Biomarker MSC-C5b-9: A Prospective, Randomized, Open-Label, Multicenter Clinical Trial
Brief Title: The Combination of ATRA and Eltrombopag as the Treatment of Steroid-resistant/Relapse ITP Based on MSC-C5b-9
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Collaborators: Beijing Friendship Hospital (Other); Beijing Tongren Hospital (Other); Beijing Hospital (Other Government); Navy General Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Xiao Hui Zhang, Vice president of Peking Univeristy Institute of Hematology, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-1-4082
Record Dates: First submitted 2022-06-25; First posted 2022-06-30 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2024-12

CONDITIONS: Purpura, Thrombocytopenic, Idiopathic
Keywords: Resistant/recurrent ITP; MSC-C5b-9 marker; all-trans retinoic acid; Eltrombopag; prospective clinical study
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Tretinoin; eltrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Eltrombopag (Active Comparator): The initial dose of eltrombopag was 50 mg/time, once a day. According to the clinical standard of eltrombopag dose adjustment in the research protocol set by the research group, the dose was increased when the platelet count was lower than 5×109/L. The highest is 75mg/d, if the dose is higher than 200×109/L, the dose is reduced. When the dose is higher than 400×109/L, the drug is temporarily discontinued, and the drug is repeated according to the platelet count. The treatment course is 12 weeks.
  Interventions: Drug: Eltrombopag
- ATRA and Eltrombopag (Experimental): ATRA 10 mg, 2 times a day, orally; The initial dose of eltrombopag was 50 mg/time, once a day. According to the clinical standard of eltrombopag dose adjustment in the research protocol set by the research group, the dose was increased when the platelet count was lower than 5×109/L. The maximum dose is 75 mg/d, the dose is reduced if it is higher than 200×109/L, and the drug is temporarily discontinued when it is higher than 400×109/L, and the drug is repeated according to the platelet count. The treatment course is 12 weeks.
  Interventions: Drug: all-trans retinoic acid; Drug: Eltrombopag

INTERVENTIONS:
Drug: all-trans retinoic acid — ATRA 10 mg, 2 times a day, orally.The treatment course is 12 weeks.
  Other Names: retinoic acid
  Arms: ATRA and Eltrombopag
Drug: Eltrombopag — The initial dose of eltrombopag is 50 mg/time, once a day, and the dose is increased when the platelet count is lower than 5×109/L, the maximum is 75 mg/d, and the dose is higher than 200×109/L. When the drug is temporarily discontinued, the drug is re-administered according to the platelet count.The treatment course is 12 weeks.
  Other Names: TPO-RA

SUMMARY:
A Prospective, Randomized, Open-Label, Multicenter Clinical Trial study to compare the efficacy and safety of ATRA plus eltrombopag compared to eltrombopag monotherapy in the treatment of steroid-resistant/relapsed immune thrombocytopenia (ITP).

DETAILED DESCRIPTION:
The investigators are undertaking a parallel group, multicenter, randomized controlled trial of patients with ITP in China. Patients were tested for MSCs, and they were divided into MSC-C5b-9+ group and MSC-C5b-9- group according to the test results, and the two groups were randomized to ATRA + eltrombopag and eltrombopag monotherapy group. Platelet count, bleeding and other symptoms were evaluated before and after treatment. Adverse events are also recorded throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* 1. Isolated thrombocytopenia (platelet count <30 × 109/L); 2. age > 18 years; 3. normal white blood cells and red blood cells on bone marrow examination; 4. increased number of megakaryocytes (bone marrow examination was performed in all patients except for myelofibrosis or other conditions that can cause thrombocytopenia disease); 5. the spleen was normal in size; 6. Eastern Cooperative Oncology Group status score (ECOG score) ≤ 2; 7. ineffective or relapsed after at least 1 course of full-dose full-course hormone therapy; 8. Failure of prior ITP therapy (eg, hormones, splenectomy, and cyclosporine) and at least 4 weeks from enrollment.

Exclusion Criteria:

* 1. Secondary ITP such as drug-related thrombocytopenia; 2. thrombocytopenia due to viral infection (HIV, hepatitis B virus, or hepatitis C virus); 3. severe cardiac, renal, hepatic, or respiratory insufficiency; 4. severe immunodeficiency; 5. pregnancy or lactation; 6. myelodysplasia or Myelofibrosis; 7. history of malignancy; 8. ongoing immunosuppressive therapy for other diseases; 9. patients previously treated with eltrombopag were excluded from this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2022-10-12 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Sustained Response Rate (SR) at 18 months | 18 months
  The maintenance of platelet count ≥ 30 x 10^9/L, at least 2-fold increase of the baseline count, the absence of bleeding, and no need for rescue medication at the 18-month follow-up

SECONDARY OUTCOMES:
Complete response rate (CR) | 18 months
  The complete response (CR) was defined as platelet count more than 100×10^9/L and absence of bleeding.
Response rate (R) | 18 months
  The Response rate (R) was defined as platelet count more than 30×10^9/L and more than 2 times higher than baseline, without bleeding
Inefficiency (NR) | 18 months
  Platelet count <30×10^9/L, or less than 2-fold increase from baseline or associated with bleeding
Recurrence rate (relapse) | 18 months
  After the treatment is effective, the platelet count drops below 30×10^9/L or drops to less than 2 times the basal value, or bleeding symptoms occur
Early response | 1 week
  Platelet count ≥30×10^9/L and at least doubling baseline at 1 wk.
Initial response | 1 month
  Initial response as platelet count more than 30×10^9/L and at least 2-fold increase of the baseline count and absence of bleeding.
Time to response (TTR) | 18 months
  The time from starting treatment to time of achievement of CR or R
Time to relapse (duration of efficacy) | 18 months
  The time from achievement of CR or R to time of relapse

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohui Zhang, MD, Principal Investigator — Study Principal Investigator Peking University People's Hospital
Locations (5):
- China (5):
  - Peking University Insititute of Hematology, Peking University People's Hospital, Beijing, Beijing Municipality
  - Beijing Tongren hospital, Beijing, Beijing Municipality
  - Department of Hematology, Beijing Friendship Hospital, Capital Medical University, Beijing
  - Department of Hematology, Beijing Hospital, Beijing
  - Department of Hematology, Senior Department of Hematology, the Fifth Medical Center of PLA General Hospital, Beijing